CLINICAL TRIAL: NCT06677476
Title: Developing and Determining the Effect of Mobile Application for Patients Who Will Have Cardiac Surgery and Cardiovascular Surgery Intensive Care Unit Nurses
Brief Title: Development of a Mobile Application and Determination of Its Effects
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Berrin Pazar, Assistant Professor, Lokman Hekim University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023103
Record Dates: First submitted 2024-10-25; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Surgery; Mobile Application; Patient Education
Keywords: Intensive care nursing; Surgery Nursing; Nursing Care; Heart surgery; Mobile application development

STUDY DESIGN:
Intervention Model Description: Training will be given on the mobile application to be downloaded to the mobile phone.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mobile application training group (Experimental): The group that will be trained by downloading the mobile application to their mobile phones
  Interventions: Other: mobile application training

INTERVENTIONS:
Other: mobile application training — Researchers compiled literature information and used their expertise to create mobile application content. This content will be downloaded to mobile phones via mobile application software and participants will be trained.

SUMMARY:
It has been determined that patients who have undergone heart surgery have a lack of knowledge about preoperative preparation and postoperative intensive care unit. In order to eliminate the lack of knowledge, patient education has gained importance in the preoperative period. At the same time, it is stated that nurses working in cardiovascular surgery intensive care units need continuous education to cope with the difficulties related to the increasing complexity of patient conditions and technology. With the advancement of technology, mobile applications have become an integral part of the continuous education of patients and nurses. This project was planned to evaluate the effect of the mobile application to be developed for patients who will undergo heart surgery on patient outcomes and the effect of the mobile application to be developed for nurses who provide patient care in intensive care units on the self-efficacy of nurses. In the first step of the project, the content of the mobile application will be developed, expert opinions will be obtained and the comprehensibility of patients and nurses will be tested. The software of the mobile application will be completed by shooting the necessary videos for the final content. In the second step of the project, the effect of the developed mobile application on anxiety, comfort and intensive care unit experiences in patients who meet the inclusion criteria will be examined. A randomized controlled experimental design will be used in this stage. State-Trait Anxiety Inventory, Early Postoperative Comfort Scale (EPQI), Intensive Care Experiences Scale will be used to collect data. Self-Efficacy Scale will be applied to nurses without randomization before and after using the mobile application. Data obtained in the study will be evaluated in a computer environment using SPSS data package program. In statistical decisions, p<0.05 level will be accepted as a significant difference indicator.

DETAILED DESCRIPTION:
Population and sample of the project:

The population will consist of all patients undergoing surgery in the Department of Cardiovascular Surgery at Lokman Hekim University Akay Hospital and treated in the ICU. Power analysis was performed to determine the number of people to be included in the study. The power of the test was calculated with the G*Power 3.1 programme. As a similar study in the relevant literature, Pehlivan (2021) calculated the effect size for the state anxiety difference as 0.646. In order to exceed the 90% value in determining the power of the study; 84 people, including 42 people in groups with a significance level of 5% and an effect size of 0.646, should be reached (df=82; t=1.664). Considering the high power of the test and the losses in the study, it was aimed to reach a total of 100 people, including 50 people in the groups.

All nurses working in the ICU of the Cardiovascular Surgery Department of Lokman Hekim University Akay Hospital will constitute the population of the study (N:10) and the nurses who volunteered to participate in the study will constitute the sample. Without randomisation for nurses, all nurses will be ensured to use the mobile application, pre-test and post-test will be performed.

Translated with DeepL.com (free version)

ELIGIBILITY:
Inclusion Criteria:

for patients;

* having elective open heart surgery,
* being a volunteer,
* being 18 years of age or older,
* knowing Turkish,
* not having a mental disability that may prevent communication,
* not having hearing or vision problems,
* having the ability to use the mobile application.

Exclusion Criteria:

* having emergency surgery,
* having previously been treated in the ICU,
* wanting to leave the study at any stage of the project.

Inclusion Criteria:

for nurses;

* working in the cardiovascular surgery ICU,
* being a volunteer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Patients' anxiety | As soon as you are admitted to the clinic and on the first day after the surgery
  The State and Trait Anxiety scale can be scored between a minimum of 20 and a maximum of 80. As the score increases, the level of anxiety increases.
blood pressure | Immediately after admission to the clinic, after waking up in the intensive care unit and on the first day after surgery
  Blood pressure will be measured manually

SECONDARY OUTCOMES:
comfort of patients | 1st day after surgery
  Early Postoperative Comfort Scale; The highest total score is 144 and the lowest total score is 24. A low score indicates poor comfort and a high score indicates good comfort.

OTHER OUTCOMES:
satisfaction with mobile application | after using the app (1st day after surgery)
  no scale will be used. Participants will be asked to evaluate the mobile application.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Meriç, assoc prof, Study Chair — Lokman Hekim University; Kaan Kaya, assoc prof, Study Director — Ankara Etlik City Hospital
Locations (1):
- Gulhane Medical Faculty, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No